CLINICAL TRIAL: NCT00128804
Title: Bioefficacy and Bioavailability of Beta-Carotene in Oil and in a Mixed Diet in Ileostomy Patients Measuring Using Specifically 13C-Labelled Beta-Carotene and Retinol
Brief Title: The STOVITA Study - Bioefficacy of Beta-Carotene in Oil and in a Mixed Diet in Ileostomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Dairy Organization (NZO) (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STOVITA-2004-03-19-NZO; NZO-2002-07
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2005-08-29 (Estimated); Status verified 2005-08

CONDITIONS: Healthy; Ileostomy
Keywords: vitamin A; beta Carotene; diet; nutrition; nutritional requirements
MeSH Terms: interventions — Absorption

INTERVENTIONS:
Behavioral: absorption and conversion of beta-carotene in human gastrointestinal (GI) tract

SUMMARY:
A controlled dietary intervention study will be carried out based on the stable isotope method the investigators have developed to quantify both the absorption of beta-carotene and its bioconversion to retinol in oil and in a mixed diet. For 4 weeks the participants will consume 2 capsules/day, 7 days/week with each capsule containing 100-mg [13C10] beta-carotene and 100-mg [13C10] retinyl palmitate. For two weeks they will consume a diet with high levels of beta-carotene in vegetables and fruits and for the other 2 weeks they will consume a diet with low levels of beta-carotene in vegetables and fruits supplemented with an extra amount of beta-carotene in oil. Samples of blood and faeces will be taken. The study hypothesis is that the absorption of beta-carotene in oil in comparison with the absorption of beta-carotene in a mixed diet differs by a factor of 3 to 6. The investigators want to measure the influence of the food matrix of vegetables and fruits on the absorption of beta-carotene in ileostomy patients on a western diet.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 75 years old
* Body mass index (BMI) between 18 and 30 kg/m2
* Willing to consume the controlled diet and not consume other food items
* Willing to consume the capsules every day
* Having a functional ileostomy (output <2 L/d)
* Relatively good medical, nutritional and health status

Exclusion Criteria:

* Diseases which disturb normal digestion and absorption
* Use of (oral) drugs suspected of interfering with fat-soluble vitamin absorption
* Excessive alcohol consumption (>30 g/d)
* Consumption of vitamin or carotenoid supplements 6 weeks before and during the study
* Not too low or high levels of serum beta-carotene and retinol
* Normal hemoglobin, hemocytometry, creatinine, ALAT, alkaline phosphatase, and cholesterol blood values (compared with laboratory references)
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2004-07; Study Completion 2004-10

PRIMARY OUTCOMES:
levels of retinol and carotenoids and the degree of isotopic enrichment in serum (fasting blood sample) and in faeces (72 hour collection) at the start and at the end of each of the 2-week periods

CONTACTS AND LOCATIONS:
Overall Officials: Ton HJ Naber, MD PhD, Study Director — Radboud University Medical Center; Clive E West, PhD DSc, Principal Investigator — Radboud University Medical Center; Carolien A Bouwman, MSc, Study Chair — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] van Lieshout M, West CE, Muhilal, Permaesih D, Wang Y, Xu X, van Breemen RB, Creemers AF, Verhoeven MA, Lugtenburg J. Bioefficacy of beta-carotene dissolved in oil studied in children in Indonesia. Am J Clin Nutr. 2001 May;73(5):949-58. doi: 10.1093/ajcn/73.5.949. PMID 11333850
- [Background] van Lieshout M, West CE, van Breemen RB. Isotopic tracer techniques for studying the bioavailability and bioefficacy of dietary carotenoids, particularly beta-carotene, in humans: a review. Am J Clin Nutr. 2003 Jan;77(1):12-28. doi: 10.1093/ajcn/77.1.12. PMID 12499318
- [Derived] Van Loo-Bouwman CA, Naber TH, van Breemen RB, Zhu D, Dicke H, Siebelink E, Hulshof PJ, Russel FG, Schaafsma G, West CE. Vitamin A equivalency and apparent absorption of beta-carotene in ileostomy subjects using a dual-isotope dilution technique. Br J Nutr. 2010 Jun;103(12):1836-43. doi: 10.1017/S0007114509993849. Epub 2010 Feb 5. PMID 20132586